CLINICAL TRIAL: NCT01986179
Title: Impact of Remote Interpreter Modality on Comprehension, Communication Quality, and Consistency of Interpreter Use in the Pediatric Emergency Department
Brief Title: Comparing Remote Interpreter Modalities in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, K. Casey Lion, Assistant Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14647
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Limited English Proficient Patients and Families

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Interpretation (Active Comparator): These families will be assigned to use telephone interpretation throughout the ED visit.
  Interventions: Other: Telephone Interpretation
- Video Interpretation (Experimental): These families will be assigned to use video interpretation throughout the ED visit.
  Interventions: Other: Video Interpretation

INTERVENTIONS:
Other: Telephone Interpretation — Professional interpretation provided over the phone by a national network of certified medical interpreters
  Arms: Telephone Interpretation
Other: Video Interpretation — Professional interpretation provided over video by a national network of certified medical interpreters
  Arms: Video Interpretation

SUMMARY:
Professional interpretation improves quality of care for patients with limited English proficiency (LEP). However, many health care settings lack access to professional interpreters, and even in locations with good access, logistical factors and perceived barriers have limited their widespread use. Remote methods of professional interpretation, including telephone and video, hold great promise for expanding access, but only limited data exist on the relative impacts of these modalities on patient care and provider uptake. Comparing how these modalities impact multiple aspects of health care quality, including family comprehension, provider communication, and consistency of provider interpreter use will inform dissemination of strategies for delivery of safe, efficient, and equitable care to LEP families.

Aim 1: To determine whether randomly assigned remote interpreter modality (telephone versus video) impacts parent-reported quality of communication and interpretation, diagnosis comprehension, and length of stay (LOS) among LEP Spanish-speaking families seen in a pediatric Emergency Department (ED).

Hypothesis 1: Parent-reported quality of communication and interpretation and parent diagnosis comprehension will be higher among families assigned to video interpretation compared to telephone interpretation.

Hypothesis 2: LOS will not differ between families assigned to video and telephone interpretation.

Aim 2: To determine whether assigned interpreter modality is associated with provider decision to communicate without professional interpretation.

Hypothesis 3: Parent-reported provider communication without professional interpretation (e.g. using the patient or a family member to interpret for some part of the visit) will be lower for families assigned to video interpretation compared to telephone interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Preferred language for medical care of Spanish
* At least one primary caregiver requires interpretation
* Presenting to Seattle Children's ED during recruiting hours

Exclusion Criteria:

* Triage level 1 (life-threatening illness)
* No parent or legal guardian present
* Reason for visit is concern for abuse
* reason for visit is primary behavioral or psychiatric complaint

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Communication Quality | Once, 1-7 days after the ED visit
  We will use the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Child Visit Survey 2.0 communication composite, which includes 5 items.
Interpretation Quality | Once, 1-7 days after ED visit
  Interpretation quality will be measured with the Interpreter Satisfaction Survey (7 items).
Diagnosis Comprehension | Once, 1-7 days after ED visit
  Parents will be asked to name their child's diagnosis. Clinician-recorded diagnosis will be obtained from chart review for comparison. Responses will be classified as correct, incorrect, or vague/incomplete, using a method we have employed previously.
Consistency of Interpreter Use | Once, 1-7 days after ED visit
  Parents will be asked to report on the frequency with which providers used each of a list of potential communication methods (e.g. telephone interpreter, family or friend, spoke in English without an interpreter present). Response options are never, sometimes, frequently, or always.

SECONDARY OUTCOMES:
Length of ED stay | Once, after ED visit
  Time from arrival in Emergency Department to discharge home or admission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: K. Casey Lion, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital Emergency Department, Seattle, Washington, United States

REFERENCES:
- [Derived] Lion KC, Gritton J, Scannell J, Brown JC, Ebel BE, Klein EJ, Mangione-Smith R. Patterns and Predictors of Professional Interpreter Use in the Pediatric Emergency Department. Pediatrics. 2021 Feb;147(2):e20193312. doi: 10.1542/peds.2019-3312. PMID 33468598
- [Derived] Lion KC, Brown JC, Ebel BE, Klein EJ, Strelitz B, Gutman CK, Hencz P, Fernandez J, Mangione-Smith R. Effect of Telephone vs Video Interpretation on Parent Comprehension, Communication, and Utilization in the Pediatric Emergency Department: A Randomized Clinical Trial. JAMA Pediatr. 2015 Dec;169(12):1117-25. doi: 10.1001/jamapediatrics.2015.2630. PMID 26501862